CLINICAL TRIAL: NCT01603537
Title: Impact of Prehospital Trauma Life Support (PHTLS) Training of Ambulance Caregivers on Outcome of Traffic Injury Victims
Brief Title: The Impact of Prehospital Trauma Life Support (PHTLS) on Outcome of Traffic Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Uppsala University Hospital (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Hans Blomberg, Medical Director of the ambulance service, Uppsala University Hospital
Other Study IDs: Dnr 2007/264
Record Dates: First submitted 2012-05-15; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Traffic Accidents
Keywords: Traumatic injuries; Prehospital Trauma Life Support; Traffic accidents
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PHTLS: The exposure is defined from the dichotomization of the probability in each event/accident that at least one of the caring ambulance crew members was PHTLS certified.
- No PHTLS: Not exposed to PHTLS

SUMMARY:
Trauma is the leading cause of death among persons below 60 years of age. It is a well-established belief that optimal treatment in the early phase after trauma has a major impact on mortality, and the implementation of specific educational programs for trauma care have been a widely adopted strategy aimed at improving the outcome. This strategy has high face validity, but the underlying evidence is poor. The Prehospital Trauma Life Support (PHTLS) program was introduced in 1983 aiming to integrate prehospital trauma care with the Advanced Trauma Life Support (ATLS) program. Approximately half a million prehospital caregivers in over 50 countries have taken the PHTLS course. It has been recognized as one of the leading educational programs for prehospital emergency trauma care. However, the scientific support for improved patient outcome from courses such as PHTLS and ATLS is limited. According to a Cochrane analysis published 2010 there is no evidence to recommend advanced life-support (ALS) training for ambulance crews. Another Cochrane analysis concerning ATLS gave similar results and a recent study indicated even worsened outcome after the implementation of ATLS. An observational study in the county of Uppsala indicated reduced mortality after the implementation of PHTLS but the estimate was uncertain due to a low overall mortality. The aim of this study is to further investigate the association between PHTLS training of ambulance crew members and the outcome in trauma patients in a larger study population. To accomplish this the investigators will use an epidemiological semi-individual design applied to all victims of traffic injury that occurred during the implementation period of the PHTLS course in Sweden (1998-2004). Four outcomes and subsets of patients will be analyzed: Mortality before hospital admission, mortality within 30 days, time to death among survivors to hospital admission and return to work among survivors to hospital discharge.

DETAILED DESCRIPTION:
Source Population: Sweden is divided in 21 administrative regions providing health care (counties). In 2004 Sweden had a population of about 9 million inhabitants with an average population density of 20 inhabitants/km2.

The Emergency Medical Service (EMS)-System: The ambulance staff in Sweden consists of registered nurses and emergency medical technician (EMT) equivalents (nursing assistants with special ambulance training).

Statistics: Hierarchical random effects models will be used to model the binary outcomes. Cox proportional hazards models to analyze the time to event outcomes. The difference in mean predicted outcome between the PHTLS group and the non-PHTLS group will be used to estimate the absolute risk reduction.

ELIGIBILITY:
Inclusion Criteria:

* Primary incident hospital admissions due to traffic accidents or
* Death due to traffic accidents

Exclusion Criteria:

* If a patient appears more than once, all but the first event will be excluded from the dataset.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study Population: Motor vehicle traffic crashes were selected using the causes of injury matrix developed by the National Center for Health Statistics, Centers for Disease Control and Prevention, USA.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-05 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Mortality before hospital admission. | Patients will be followed up to death or at least one year after inclusion.
  Injury deaths not associated with a hospital admission.
Mortality within 30 days. | Patients will be followed up to death or at least one year after inclusion.
  Deaths within 30 days including all deaths, prehospital and hospital, up to 30 days from the injury event.
Time to death among survivors to hospital admission. | Patients will be followed up to death or at least one year after inclusion.
  Time to death among patients associated with a hospital admission.
Return to work among survivors to hospital discharge. | Patients will be followed up to occured event or at least one year after inclusion.
  Number of patients returned to work per time-unit of observation after the injury event among all patients discharged from hospital, not dead, and that was working before the accident.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Gedeborg, PhD, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, County of Uppsala, Sweden

REFERENCES:
- [Background] Krug EG, Sharma GK, Lozano R. The global burden of injuries. Am J Public Health. 2000 Apr;90(4):523-6. doi: 10.2105/ajph.90.4.523. PMID 10754963
- [Background] Trunkey DD, Lim RC Jr, Blaisdell FW. Traumatic injury. A health care crisis. West J Med. 1974 Jan;120(1):92-4. No abstract available. PMID 4812216
- [Background] Collicott PE, Hughes I. Training in advanced trauma life support. JAMA. 1980 Mar 21;243(11):1156-9. PMID 7359667
- [Background] Jayaraman S, Sethi D. Advanced trauma life support training for ambulance crews. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD003109. doi: 10.1002/14651858.CD003109.pub2. PMID 20091538
- [Background] Jayaraman S, Sethi D. Advanced trauma life support training for hospital staff. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD004173. doi: 10.1002/14651858.CD004173.pub3. PMID 19370594
- [Background] Drimousis PG, Theodorou D, Toutouzas K, Stergiopoulos S, Delicha EM, Giannopoulos P, Larentzakis A, Katsaragakis S. Advanced Trauma Life Support certified physicians in a non trauma system setting: is it enough? Resuscitation. 2011 Feb;82(2):180-4. doi: 10.1016/j.resuscitation.2010.10.005. Epub 2010 Nov 30. PMID 21122975
- [Background] Johansson J, Blomberg H, Svennblad B, Wernroth L, Melhus H, Byberg L, Michaelsson K, Karlsten R, Gedeborg R. Prehospital Trauma Life Support (PHTLS) training of ambulance caregivers and impact on survival of trauma victims. Resuscitation. 2012 Oct;83(10):1259-64. doi: 10.1016/j.resuscitation.2012.02.018. Epub 2012 Feb 23. PMID 22366502
- [Background] Recommended framework for presenting injury mortality data. MMWR Recomm Rep. 1997 Aug 29;46(RR-14):1-30. PMID 9301976